CLINICAL TRIAL: NCT06932497
Title: Gemelli Longitudinal Cohort on Long-term Outcomes in RheumatIc diseAses
Acronym: GLORIA
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 7235
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Rheumatic Disease
MeSH Terms: conditions — Rheumatic Diseases | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples Without DNA — Outcome predictors for GLORIA will be selected from variables routinely collected according to clinical care. The main predictors will include.
  * Laboratory Variables: derived as per clinical practice from blood, synovial fluid, bronchoalveolar lavage, urine, and feces
  * Histological Data: derived from biopsies performed as per clinical practice, involving joints, enthesis, skin, muscle, salivary glands, lungs, and gastrointestinal tract.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rheumatic diseases: Enrolled patients must be older than 18 years and present at least one of the following:
  * A clinically defined diagnosis of immune-mediated CRD (primary arthritis, vasculitis, connective tissue disease, or auto-inflammatory syndromes).
  * A clinically defined diagnosis of degenerative or metabolic CRD (osteoarthritis, crystal-induced arthritis, osteoporosis, articular disease associated with endocrine or metabolic diseases)
  * A clinically defined diagnosis of FM.
  * Undifferentiated CRD-related conditions at high risk of clinical evolution (Inflammatory joint pain with auto-antibody positivity or personal/family history of psoriasis, Raynaud's phenomenon, sicca syndrome or photo-sensibility with auto-antibody positivity, interstitial lung disease with auto-antibody positivity, uncomplicated osteopenia).
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Standard of care — Standard of care according to national and international guideline or recommendations

SUMMARY:
Chronic rheumatic diseases (CRDs) are major determinant of disability in the general population. Particularly, immune-mediated CRDs also represent a significant cause of morbidity and mortality among younger individuals. CRDs lead to substantial direct costs related to healthcare service use and pharmacological expenses, as well as indirect social costs. Proper prognostic stratification of CRD patients could tailor diagnostic and therapeutic interventions to improve clinical outcomes and strategically allocate healthcare resources while minimizing both direct and indirect costs.

Reported prognostic predictors in CRDs are largely derived from randomized therapeutic trials and therefore mostly reflect short-term outcomes under controlled experimental conditions. A real-life research could provide crucial information about long-term outcomes including survival, impact of comorbidities and polypharmacotherapy, and inform on healthcare costs.

The Gemelli longitudinal cohort on Long-term Outcomes in Rheumatic Diseases (GLORIA) aims to define shared and disease-specific predictors of long-term disability, organ damage, mortality, and healthcare costs for patients under the care of the Division of Rheumatology at the Fondazione Policlinico Universitario A. Gemelli IRCCS - Catholic University of the Sacred Heart in Rome. This study will adopt an electronic database identified for collecting and analyze data (REDcap Research Electronic Data Capture platform), compliant with general data protection regulation (GDPR) law.

Predictors will be selected from routinely collected demographic, clinical, laboratory, histological, and instrumental data. Additional blood samples may be collected from newly diagnosed patients or when diagnostic or therapeutic interventions are required according to clinical practice. Excepted for additional collection of peripheral blood, no additional procedure will be therefore performed.

DETAILED DESCRIPTION:
Rationale of GLORIA Chronic rheumatic diseases (CRDs) represent a heterogeneous group of conditions with varying epidemiological, pathophysiological, and clinical aspects. CRDs are characterized substantial impact on population morbidity and mortality and relevance in terms of public health decision making and social costs. A timely and accurate definition of the prognosis for CRDs patients is crucial for improving clinical outcomes, as well as for strategically allocating healthcare resources and minimizing indirect economic and non-economic costs.

The most significant CRDs in terms of prevalence or need for intensive care fall into three main categories: autoimmune and inflammatory immune-mediated diseases, metabolic and degenerative diseases, and extra articular pain syndromes of which fibromyalgia (FM) is the most diffuse.

The category of autoimmune or inflammatory immune-mediated diseases includes conditions attributed to aberrant activation of the immune system, with the highest prevalence conditions being primary arthritis and conditions that are individually less common but collectively epidemiologically relevant such as connective tissue diseases, vasculitis, and autoinflammatory syndromes. Similarly to organ-specific autoimmune conditions, these have shown an increasing incidence in the last decades. Most of them are associated with multi-organ involvement and potentially life-threatening complications.

Degenerative and metabolic pathologies include primary and secondary osteoarthritis, crystal arthropathies, and metabolic bone diseases, with osteoporosis and algodystrophy being the most prevalent forms. These conditions are extensively associated with aging processes and endocrine-metabolic diseases. Their prevalence has increased over the last decades considering the demographic trends of the Italian population and concurrently with the rising incidence of closely related conditions such as the so called "metabolic syndrome". They represent a relevant morbidity burden in the general population around the world and their complications have been associated with increased mortality.

Finally, FM is the most common cause of chronic widespread musculoskeletal pain particularly in women between 20 and 55 years of age. FM is often accompanied by fatigue, cognitive disorders, psychiatric symptoms, and multiple somatic symptoms. It is characterized by forms of central sensitization in the absence of documented inflammation affecting joints, muscles, ligaments, and tendons.

ELIGIBILITY:
Minimum Age: 18 Years Sex: All Gender Based:No

Inclusion criteria:

* sign an informed consent
* A clinically defined diagnosis of immune-mediated CRD (primary arthritis, vasculitis, connective tissue disease, or auto-inflammatory syndromes).
* A clinically defined diagnosis of degenerative or metabolic CRD (osteoarthritis, crystal-induced arthritis, osteoporosis, articular disease associated with endocrine or metabolic diseases)
* A clinically defined diagnosis of FM.
* Undifferentiated CRD-related conditions at high risk of clinical evolution (Inflammatory joint pain with auto-antibody positivity or personal/family history of psoriasis, Raynaud's phenomenon, sicca syndrome or photo-sensibility with auto-antibody positivity, interstitial lung disease with auto-antibody positivity, uncomplicated osteopenia).

Exclusion criteria:

- Active follow-up and inability to express informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with chronic rheumatic diseases.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2030-04-07 (Estimated); Study Completion 2035-04-07 (Estimated)

PRIMARY OUTCOMES:
HAQ-DI | 10 years
  Degree of disability in CRD patients, quantified according to the Health Assessment Questionnaire-Disability Index.

SECONDARY OUTCOMES:
Mortality | 10 years
  CRD-related mortality and mortality from any cause.
Complications | 10 years
  Major disease- or treatment-related complications, such as severe infections, cancer, major cardiovascular events, bone fractures, and organ failure.
Heathcare service access | 10 years
  Access to outpatient clinics, day hospitals, emergency services, and hospital wards, along with related healthcare costs.
Drug and surgery access | 10 years
  Access to medications and surgical procedures, and their associated healthcare costs.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Antonietta D'Agostino, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: No